CLINICAL TRIAL: NCT01890369
Title: Modulation of Muscle Protein Metabolism by Essential Amino Acids
Acronym: Aj1B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: Ajinomoto Co., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: B13122012 GEM BMS
Record Dates: First submitted 2013-06-26; First posted 2013-07-01 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Old Age
Keywords: Old Age; Sarcopenia; Amino Acid; Muscle
MeSH Terms: conditions — Sarcopenia | interventions — Leucine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Early leucine refeed (Experimental): 15g Mixed Essential Amino Acids. 90 min delay. 3g Leucine
  Interventions: Dietary Supplement: 15g Mixed Essential Amino Acids; Dietary Supplement: 3g Leucine
- Early EAA refeed (Experimental): 15g Mixed Essential Amino Acids. 90 min delay. 15g Mixed Essential Amino Acid REFEED
  Interventions: Dietary Supplement: 15g Mixed Essential Amino Acids; Dietary Supplement: 15g Mixed Essential Amino Acid REFEED
- Mid latency EAA refeed (Experimental): 15g Mixed Essential Amino Acids. 150 min delay. 15g Mixed Essential Amino Acid REFEED
  Interventions: Dietary Supplement: 15g Mixed Essential Amino Acids; Dietary Supplement: 15g Mixed Essential Amino Acid REFEED
- Late latency EAA refeed (Experimental): 15g Mixed Essential Amino Acids. 210 min delay. 15g Mixed Essential Amino Acid REFEED
  Interventions: Dietary Supplement: 15g Mixed Essential Amino Acids; Dietary Supplement: 15g Mixed Essential Amino Acid REFEED

INTERVENTIONS:
Dietary Supplement: 15g Mixed Essential Amino Acids — Dissolved in 250ml water.
Dietary Supplement: 3g Leucine — Dissolved in 250ml water.
  Arms: Early leucine refeed
Dietary Supplement: 15g Mixed Essential Amino Acid REFEED — Dissolved in 250ml water.
  Arms: Early EAA refeed; Late latency EAA refeed; Mid latency EAA refeed

SUMMARY:
The investigators plan to explore the ability of amino acids, the building blocks of proteins in our bodies and in the food we eat, to stimulate muscles to grow and stay strong. The investigators will investigate how rapidly after one meal the human body is ready to make use of a second meal and look at the molecular mechanisms underlying this. The investigators will look at these phenomena in older men as this group is known to be subject to a gradual loss of muscle mass and strength.

DETAILED DESCRIPTION:
Muscles can stay very constant in size for much of adult life yet dramatic wasting is seen in advanced age and ill health. A better understanding of how muscles regulate their size will help design treatments to slow wasting in disease and to promote active aging. We plan to study a group of older men, ~70yrs, the age at which muscle bulk starts to decrease, to observe how the muscles respond to feeding. We will provide a drink that contains the digested products of proteins from which muscles are built. Taking blood samples and some tiny biopsies of muscle (done under local anaesthesia) will allow us to measure muscle turnover and we will be able to measure for how long after a meal muscles actively take in nutrients before becoming "full". We will also measure how long the muscle remains "full" before it returns to a state where it can again be stimulated to take in nutrients. We will also explore if leucine, one of the component parts of protein (especially in meat and dairy products) and a food widely used supplement, can promote the early re-stimulation of muscle by eating.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 65-75yrs
* BMI 18-28

Exclusion Criteria:

* Type 2 Diabetes mellitus
* Neurological Disease
* Significant cardiac, hepatic or renal disease
* Active malignancy
* Medication inc. Corticosteroids, NSAID use, Beta adrenoblockers.

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Myofibrillar Fractional Synthetic Rate | 6-10hrs
  Assessed by gas-chromatography-combustion-mass spectrometry, using incorporation of a stable isotope tracer (13-C-6 Phe)

SECONDARY OUTCOMES:
Leg blood flow | 6-10hrs
  Common femoral bulk flow (Doppler USS)
mTORC1 and AKT phosphorylation | 6-10hrs
  Western Immunoblotting
Muscle Protein Breakdown | 6-10hrs
  By Arteriovenous limb balance

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Atherton, PhD, Principal Investigator — University of Nottingham
Locations (1):
- School of Graduate Entry Medicine, Derby, United Kingdom